CLINICAL TRIAL: NCT05488379
Title: Well Child Care Intervention for Infants of Mothers in Treatment for Opioid Use Disorder
Brief Title: Child Healthcare at MATER - Pediatric Study
Acronym: CHAMPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Alfred I. duPont Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17540
Record Dates: First submitted 2022-04-01; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Opioid Use Disorder
Keywords: Group well child care; Child developement; Parenting behavior; Healthcare quality; Healthcare experience
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual well child care (No Intervention): Individuals randomized to the control arm will receive routine individualized well child care after birth hospital discharge.
- Group well child care (Experimental): Individuals randomized to the intervention arm will participate in group well child care after birth hospital discharge.
  Interventions: Other: Group well child care

INTERVENTIONS:
Other: Group well child care — Beginning with the 1-month well child care visit, mother-infant dyads will participate in well child care together, with subsequent visits occurring at the American Academy of Pediatrics recommended intervals (2, 4, 6, 9, 12, 15, and 18 months of age).
  Other Names: CenteringParenting
  Arms: Group well child care

SUMMARY:
The objective of this project is to implement and evaluate a group model of well child care for mothers in treatment for opioid use disorder and their children that addresses the specific health needs and concerns of opioid-exposed infants, is trauma informed, and is embedded within a maternal opioid use disorder treatment program. 108 mother-infant dyads will be randomized 1:1 to group well child care or individual well child care, and followed over an 18 month period. Qualitative and quantitative data will be collected at multiple time points. The efficacy of group well child care to improve health and healthcare-related outcomes will be evaluated.

DETAILED DESCRIPTION:
This is a single-site cluster randomized controlled trial. Over an 18-month period, 108 pregnant women receiving treatment for opioid use disorder will be identified, screened, and enrolled into the study. Beginning with the birthdate of the first infant born in the study, 18 consecutive 1-month birth intervals will be randomized in a 1:1 ratio to one of two study arms: (1) group well child care or (2) individual well child care. Nine birth clusters will be randomized to individual well child care(control arm) and nine birth clusters will be randomized to group well child care(intervention arm), with concealment of randomization from enrolled participants until they give birth. All study participants will be included in the study until their child is approximately 18 months of age. All study participants will have a total of 5 assessment visits with research personnel; visits will occur immediately following enrollment into the study (baseline), prior to the participant's child turning 1 month of age, and within 4 weeks of the participant's child turning 6, 12, and 18 months of age. The efficacy of group well child care to improve health and healthcare-related outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* at least 28 weeks pregnant or less than 2 weeks postpartum
* receiving treatment for opioid use disorder
* ability to read and speak English
* plans to parent infant after delivery
* intent to seek pediatric care within Nemours/Thomas Jefferson University system
* intent to remain in the Philadelphia area for the next 2 years

Exclusion Criteria:

* inability to speak English
* plans to move outside of the Philadelphia area in the next 2 years
* plans to not parent infant after delivery
* plans to seek pediatric care outside of the Nemours/Thomas Jefferson University System

Following a live birth, participants will remain eligible to continue in the study unless the mother or infant experiences the following: gestational age at time of delivery less than or equal to 32 weeks or illness or clinical complication warranting prolonged hospitalization after delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Well child care engagement | 18 months post-delivery
  Measured as both utilization and experience of well child care. Utilization will be defined as total number of well child care visits during the child's first 18 months of life. Adequacy of well child care during this time period will be dichotomized as adequate (7 well child care visits) or inadequate (<7 well child care visits). This definition is adapted from the Health Plan Employer Data and Information Set (HEDIS) measure for well child care. The Promoting Healthy Development Survey (PHDS) will be used to evaluate participants' perceptions of their child's well child care, including anticipatory guidance, developmental surveillance, family-centeredness, family risk assessment, and helpfulness of care.
Parenting Knowledge | 18 months post-delivery
  A survey instrument will include investigator-developed questions as well as questions from the Knowledge of Infant Development Inventory (KIDI).
Maternal-child interaction quality | 18 months post-delivery
  This will be directly assessed using a video recorded mother/child free play at 18 months. Interactions will be coded by using the Keys to Interactive Parenting Scale (KIPS). KIPS is a structured observational measure and assesses 12 domains of parenting. The domains are scored on a 1 to 5-point scale with higher scores indicating higher quality parenting behaviors.

SECONDARY OUTCOMES:
Infant healthcare utilization | 18 months of age
  lead screening; up-to-date immunization status based on the CDC immunization schedule; maternal depression screening; PEDS developmental screening; infant Hepatitis C screening among those with perinatal Hepatitis C exposure; number of acute primary care visits (sick visits); emergency department utilization and hospitalization; subspecialist referrals and visits; early intervention referral and enrollment.
Infant development | 6 months of age
  self reported using Ages & Stages Questionnaires, 3rd Edition (ASQ-3), a set of 40-item parent-reported age-specific development screening questions assessing communication, gross motor, fine motor, problem solving and personal-social skills. Scores for each of the five domains range from 0-60 with higher scores indicating typical development.
Infant development | 12 months of age
  self reported using Ages & Stages Questionnaires, 3rd Edition (ASQ-3), a set of 40-item parent-reported age-specific development screening questions assessing communication, gross motor, fine motor, problem solving and personal-social skills. Scores for each of the five domains range from 0-60 with higher scores indicating typical development.
Infant development | 18 months of age
  self reported using Ages & Stages Questionnaires, 3rd Edition (ASQ-3), a set of 40-item parent-reported age-specific development screening questions assessing communication, gross motor, fine motor, problem solving and personal-social skills. Scores for each of the five domains range from 0-60 with higher scores indicating typical development.
Maternal health behaviors | 12 months of age
  self-reported duration of breastfeeding, infant sleep positioning, contraception use , and repeat pregnancy.
Maternal psychosocial | 18 months of age
  depression using the Edinburgh Postnatal Depression Scale
  The EPDS is a 10-item self report used to measure postpartum depression. Scores range from 0-30, with a higher score indicating a greater severity of depression.
Maternal psychosocial | 18 months of age
  General stress using the Perceived Stress Scale (PSS; higher scores indicate higher stress)
  The Perceived Stress Scale (PSS) is a 10-item scale to measure stress. Scores range from 0-40, with higher scores indicating greater perceived stress.
Maternal psychosocial | 18 months of age
  Parenting stress using the Parenting Stress Index (PSI)
  The Parenting Stress Index (PSI) is a 36-item questionnaire assessing parental stress. Total scores range from 36 to 180, with higher scores indicating greater parental stress.
Maternal psychosocial | 18 months of age
  Social support using the Social Provisions Scale (SPS)
  The Social Provisions Scale (SPS) is one of the most frequently used scales on social support, and is validated to measure the components of social support that directly impact health outcomes: attachment, social integration, reassurance of worth, reliable alliance, guidance, and opportunity for nurturance.
Maternal return to illicit substance abuse | 18 months of age
  Any number of positive urine drug screens for illicit substance(s)
Maternal sensitivity/responsiveness | 12 months of age
  Self-reported using the Maternal Responsiveness Questionnaire, which measures the extent to which mothers respond promptly to their infants across different situations. The measure yields 3 subscales: responsiveness, non-responsiveness, and delayed responsiveness. Higher scores indicate higher tendency for responsiveness, non-responsiveness, and delayed responsiveness.
Maternal sensitivity/responsiveness | 18 months of age
  Self-reported using the Coping with Toddlers' Negative Emotions Scale (CTNES) which measures the degree to which mother perceive themselves as reactive to their children's negative affect in distressful situations.
  The CTNES consists of scenarios in which youth may experience negative emotion. Parents are asked to identify how they would respond to each scenario. Each scenario has six responses which parents rate on a 7 point Likert-scale regarding their likelihood of responding that way (1 = very unlikely, 7 = very likely). This measure has six subscales which include emotion focused, problem-focused, minimization, punitive, expressive encouragement, and distress responses. Higher scores indicate a higher presence of that parenting response.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Short, PhD, Principal Investigator — Thomas Jefferson University; Neera Goyal, MD, Principal Investigator — Nemours Al DuPont Pediatrics
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Short VL, Abatemarco DJ, Sood E, Hand DJ, Gannon M, Hossain J, Goyal NK. The Child Healthcare at MATER Pediatric Study (CHAMPS): a 2-arm cluster randomized control trial of group well child care for mothers in treatment for opioid use disorder and their children. Trials. 2023 May 17;24(1):333. doi: 10.1186/s13063-023-07357-2. PMID 37194074